CLINICAL TRIAL: NCT01266226
Title: Effect of Autologous Plasma (ACP) on Surgical Repair of Rotator Cuff Tears
Brief Title: Effect of ACP on Surgical Repair of Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Matthias Flury, Principal Investigator, Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACP01; KEK-ZH-Nr. 2010-0309/4 (Other: Regional Ethics Committee of Zurich)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff tears; ACP
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACP treated (Experimental): The patients are going to get an injection of 4mL autologous conditioned plasma under the footprint following an arthroscopic repair of the rotator cuff.
  Interventions: Device: Autologous conditioned plasma
- Control group (Placebo Comparator): The patients are going to get an injection of 4mL saline solution under the footprint following an arthroscopic repair of the rotator cuff.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Autologous conditioned plasma — 4mL autologous conditioned plasma application under the footprint following an arthroscopic repair of the rotator cuff.
  Other Names: ACP Arthrex
  Arms: ACP treated
Device: Control group — 4mL saline application under the footprint following an arthroscopic repair of the rotator cuff.
  Other Names: ACP Arthrex
  Arms: Control group

SUMMARY:
The purpose of this study is to determine if autologous plasma (ACP) is beneficial for better and faster healing following an arthroscopic repair of the rotator cuff.

DETAILED DESCRIPTION:
The shoulder joint, specially the rotator cuff, is one of the most complicated joints of the human body. If the tendon has to be fixed at the bone during surgery, the weak point in obtaining a successful surgery is the fixation of the tendon at the bone insertion site. Tendon belongs to the bradytrophic tissue conditional on the reduced blood flow, deep mitosis rate and lowered healing potential. We can boost the healing process with a selective use of PRP (platelet rich plasma). In this process, the healing site is delivered with an elevated concentration of thrombocytes and also growth factors which are constituent parts of them.

In this study, we will test the Arthrex® Double Syringe System. With this system it is possible to obtain ACP (Autologous conditioned plasma) in one centrifugation step. The supernatant contains a concentration of thrombocytes which is twice as high as in the native blood. The concentration of the growth factors is 5-25x higher according to this.

We also want to test if one application of ACP is enough to get a short- and long-term benefit in healing following a rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic rotator cuff reconstructions of degenerative or traumatic full thickness rotator cuff tears (supraspinatus and/or infraspinatus tendon) performed by Dr. Flury and Dr. Schwyzer
* Suture bridge technique
* No pregnancy at the date of the surgery for women of childbearing potential
* Signed consent form

Exclusion Criteria:

* Partial reconstruction of the rotator cuff (PASTA)
* Open reconstruction
* Tendon transfer (latissimus dorsi or pectoralis major)
* Revision surgery
* Omarthrosis (Level ≥ 2 Samilson & Prieto)
* Systemic arthritis
* Rheumatoid arthritis
* Diabetes (insulin treated)
* Requiring surgery in reconstruction of the subscapularis tendon
* Progressive fat inclusion (fatty infiltration of the rotator cuff musculature Goutallier level IV
* Acute or chronic infection
* Pathological bone metabolism
* Insufficient perfusion in the affected arm
* Neuromuscular disease in the affected arm
* Non compliance of the patient
* Disorders which handicap or inhibit the patient to follow the orders of the clinical testers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 3mo (6mo/24mo)
  The Oxford Shoulder Score used after 3 months is the primary parameter. The Score tests the ability to participate in the patients' normal life before they got injured.

SECONDARY OUTCOMES:
VAS Pain | 10d po
QuickDASH | 3/6/24mo
EQ-5D | 3/6/24 mo
ROM | 3/6/24mo
Measurement of the abduction strength | 3/6/24 mo
ASES Score | 3/6/24mo
Constant Murley Score | 3/6/24 mo
MRI/X-Ray/Ultrasonic Diagnostics | 6/24 mo
Measurement of the external rotation strenght | 3/6/24 mo

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Flury, Dr, Principal Investigator — Upper Extremities Department
Locations (1):
- Schulthess Klinik, Zurich, Canton Zürich, Switzerland

REFERENCES:
- [Derived] Flury M, Rickenbacher D, Schwyzer HK, Jung C, Schneider MM, Stahnke K, Goldhahn J, Audige L. Does Pure Platelet-Rich Plasma Affect Postoperative Clinical Outcomes After Arthroscopic Rotator Cuff Repair? A Randomized Controlled Trial. Am J Sports Med. 2016 Aug;44(8):2136-46. doi: 10.1177/0363546516645518. Epub 2016 May 16. PMID 27184542